CLINICAL TRIAL: NCT02493010
Title: Arousal Detection and Training for Social Anxiety Disorder (SAD)
Brief Title: Arousal Training for Social Anxiety Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke-NUS Graduate Medical School (Other)
Collaborators: Agency for Science, Technology and Research (Other); Singapore General Hospital (Other)
Responsible Party: Principal Investigator, Lee Tih Shih, Associate Professor, Duke-NUS Graduate Medical School
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: B-14-098
Record Dates: First submitted 2014-07-24; First posted 2015-07-09 (Estimated); Last update posted 2017-12-19 (Actual); Status verified 2017-12

CONDITIONS: Social Anxiety
Keywords: Virtual Reality Exposure Therapy; Computerized Cognitive Behavioral Therapy; Public Speaking; Social Phobia; Biofeedback
MeSH Terms: conditions — Speech; Phobia, Social

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Participants will undergo a 4-week intervention (once per week, 1 hour each session). Each intervention session consists of approximately 30 minutes of computerized cognitive behavioral therapy, and 30 minutes of Virtual Reality Exposure Therapy with our novel arousal-based biofeedback system. For Virtual Reality Exposure Therapy, the physiological variables of participants will be continuously monitored and presented to them as feedback. Participants will have to deliver speeches to videotaped audiences while striving to regulate their physiological arousal.
  Interventions: Device: Arousal-based biofeedback system
- Waitlist Control (No Intervention): Participants in Waitlist Control will receive no intervention in the first 4 weeks of the study. After the Intervention group has completed treatment, participants in the Waitlist Control will then undergo the same intervention as the Intervention group.

INTERVENTIONS:
Device: Arousal-based biofeedback system
  Arms: Intervention

SUMMARY:
The primary objective of the study is to examine the safety, usability and preliminary efficacy of a novel arousal-based biofeedback system in alleviating social anxiety. The investigators hypothesize that after 4 weeks of hour-long interventions, participants will show reductions pre- and post-intervention in their Liebowitz Social Anxiety Scale scores.

DETAILED DESCRIPTION:
The investigators plan to conduct a waitlist control trial.

Intervention consists of a combination of computerized cognitive behavioral therapy and arousal-based Virtual Reality Exposure Therapy. During the latter component, the physiological variables of participants, such as pulse rate and EEG, will be continuously monitored and presented as feedback to them. Participants will have to deliver speeches to videotaped audiences while striving to regulate their physiological arousal.

ELIGIBILITY:
Inclusion Criteria:

* Literate in English
* Computer literate
* Able to travel independently
* Agreeable to being video-recorded when going through study protocol
* Liebowitz Social Anxiety Scale score of 31 or more
* Public Speaking Anxiety Scale score of 60 or more
* Alcohol Use Disorders Identification Test (AUDIT) of 8 and below

Exclusion Criteria:

* Has gross visual or hearing impairments
* Has irregular heart rhythm
* On any psychoactive medication
* Involved in any other long-term research study
* Current or previous history of neuropsychiatric disorders (other than depression, which will be assessed by BDI-II)
* Suicide ideation
* Concurrent psychotherapy for any disorder
* Non-responding to a previous psychotherapy

Ages: 21 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Change in Liebowitz Social Anxiety Scale scores from Week 0 to Week 5 | Week 0 (Pre-intervention) and Week 5 (Post-intervention)
  A validated 24-item scale that is commonly used in social anxiety studies.
Satisfaction and Immersion Questionnaire | Week 4 (post-intervention) for Intervention group and Week 9 (post-intervention) for Waitlist Control group
  A 22-item questionnaire that examines how effective, enjoyable and realistic the intervention is to participants.
Safety Measure: After each intervention session (once a week), participants will be queried on whether they have experienced any physical or psychological adverse events during the study | Week 1 to Week 4 for Intervention and Week 6 to Week 9 for Waitlist Control
  The total number and severity rating of all adverse events reported will be collated at the end of the study.

SECONDARY OUTCOMES:
Change in Fear of Negative Evaluation-Brief (FNE-B) scores | Week 0 (pre-intervention) and Week 5 (post-intervention)
  According to the American Psychiatric Association's Diagnostic and Statistical Manual of Mental Disorders 5th edition (DSM-V), fear of negative evaluation is at the core of Social Anxiety Disorder. This 12-item self-report scale is a commonly used outcome measure in social anxiety studies.
Change in Self-Statements during Public Speaking (SSPS) scores | Week 0 (pre-intervention) and Week 5 (post-intervention)
  A 10-item Likert-scale instrument measuring extent of negative and positive thoughts about oneself during public speaking.
Change in Public Speaking Anxiety Scale scores from Week 0 to Week 5 | Week 0 (pre-intervention) and Week 5 (post-intervention)
  A 17-item self-rating scale that measures public speaking anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Tih-Shih Lee, MD PHD, Principal Investigator — Duke-NUS Graduate Medical School
Locations (1):
- Duke-NUS Graduate Medical School, Singapore, Singapore

REFERENCES:
- [Derived] Lin XB, Lee TS, Cheung YB, Ling J, Poon SH, Lim L, Zhang HH, Chin ZY, Wang CC, Krishnan R, Guan C. Exposure Therapy With Personalized Real-Time Arousal Detection and Feedback to Alleviate Social Anxiety Symptoms in an Analogue Adult Sample: Pilot Proof-of-Concept Randomized Controlled Trial. JMIR Ment Health. 2019 Jun 14;6(6):e13869. doi: 10.2196/13869. PMID 31199347